CLINICAL TRIAL: NCT04630405
Title: Inhaled Allergen Challenge Methodology: Assessment of SOLO Vibrating Mesh Nebulizer for Allergen-Induced Late Asthmatic Responses
Brief Title: Assessment of SOLO Vibrating Mesh Nebulizer for Allergen-Induced Late Asthmatic Responses
Acronym: SOLO-LAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Gail Gauvreau, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: McMaster-SOLO-LAR
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wright jet nebulizer (Active Comparator): Will employ the Wright jet nebulizer for use in an allergen challenge triad
  Interventions: Device: Wright jet nebulizer
- Solo vibrating mesh nebulizer (Active Comparator): Will employ the Aerogen Solo vibrating mesh device for use in an allergen challenge triad
  Interventions: Device: Aerogen Solo

INTERVENTIONS:
Device: Wright jet nebulizer — Roxon Medi-Tech, Montreal, QC, Canada
  Arms: Wright jet nebulizer
Device: Aerogen Solo — Aerogen Ltd., Galway, Ireland
  Arms: Solo vibrating mesh nebulizer

SUMMARY:
This is a mechanistic study. Having established safety with the Solo® nebulizer and the ability to predict allergen PD20 using the methacholine PD20 and STE, the current study will assess the use of the Solo® vibrating mesh nebulizer on development of allergen-induced endpoints during the late phase response.

DETAILED DESCRIPTION:
Ten asthmatic subjects (>18 years, both sexes) who have stable asthma will be recruited to undergo inhaled allergen and diluent challenges for a randomized, 2-way crossover study. The primary objective is to compare the development of LAR between allergen (known to cause EAR and LAR) and diluent control challenges (does not cause EAR and LAR) using the Solo® vibrating mesh nebulizer using a standardized inhaled allergen challenge. Subject will undergo an allergen challenge with the Solo® compared to two different controls; diluent inhalation (a negative control with saline inhalation that does not cause LAR), and versus allergen challenge with control Wright nebulizer (positive control using a nebulizer that is known to cause LAR). Up to 2 academic centres will participate in this study. The results of this study will examine if the Solo® vibrating mesh nebulizer is an adequate substitution for the Wright nebulizer.

Screening

Skin Prick test and Skin Prick test endpoint

Randomization

The washout time after each allergen/diluent challenge triad will be 3-5 weeks.

Wright Nebulizer Allergen Inhalation triad will be conducted over 3 consecutive days.

On day 1: Wright® MCT to determine methacholine PC20 for 1) eligibility, and 2) to calculate the predicted Wright® allergen PC20. If the participant meets eligibility criterion, they will undergo blood draw, sputum induction and breath analysis to measure baseline airway inflammation. Day 2: Wright® allergen challenge will be performed. Participants that demonstrate early asthmatic response (≥20% drop in FEV1 during the period10 min-2h post-allergen) and the late asthmatic response (≥15% drop in FEV1 during the period 3-7h post-allergen challenge) will be eligible to continue in the study. If the participant meets eligibility criterion, they will undergo blood draw, sputum induction and breath analysis to measure airway inflammation at 7h post-challenge. Day 3:Wright® MCT to determine the degree of allergen-induced airway hyperresponsiveness, and they will undergo blood draw, sputum induction and breath analysis to measure airway inflammation at 24h post-challenge.

The order of the Solo® nebulizer allergen and diluent challenges will be conducted in a random order during the second and third triads. These challenge triads will be conducted over 3 consecutive days. Day 1: Solo® MCT to determine methacholine PD20 to calculate the predicted Solo® allergen PD20, followed by sputum induction to measure baseline airway inflammation. Day 2: Solo® allergen challenge or diluent challenge will be performed. Sputum induction will be conducted to measure airway inflammation at 7h post-challenge. Day 3: Solo® MCT to determine the degree of airway hyperresponsiveness at 24h post-allergen and post-diluent challenge, followed by sputum induction to measure airway inflammation at 24h post-challenge.

ELIGIBILITY:
Inclusion Criteria:

* baseline FEV1 greater than or equal to 70%
* positive response to inhaled methacholine (i.e. PD20 less than 400mcg)
* evidence of atopy (i.e. positive skin prick test to an allergen that can be used for the inhalation challenge
* absence of respiratory infection for at least 4 weeks
* absence of allergen exposure (or other trigger of upper or lower respiratory symptoms) for at least 4 weeks
* current nonsmoker (ex-smoker allowed; case by case basis; investigator discretion)
* require only infrequent short-acting beta2 agonist (i.e. salbutamol or terbutaline) to treat/control asthma (i.e. no inhaled corticosteroid or combination therapies, no intranasal corticosteroid; anti-histamines etc.)
* general good health with no other medical condition, medication use or lifestyle activities that would influence the outcome of the allergen challenge
* development of allergen-induced early and late asthmatic responses

Exclusion Criteria:

* pregnant or lactating

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Development of LAR after Allergen Challenge | Basline
  The primary objective is to compare the development of LAR between allergen (known to cause EAR and LAR) and diluent control challenges (does not cause EAR and LAR) using the Solo® vibrating mesh nebulizer using a standardized inhaled allergen challenge.

SECONDARY OUTCOMES:
Development of LAR between Allergen and Diluent | based on baseline methacholine challenge and skin test endpoint results
  To compare the late asthmatic response (LAR) between inhaled allergen and inhaled diluent using the Solo® vibrating mesh nebulizer; and
Magnitude of Airway Inflammation | based on baseline methacholine challenge and skin test endpoint results
  To compare the magnitude of airway inflammation after inhaled allergen and inhaled diluent using the Solo® vibrating mesh nebulizer; and after inhaled allergen between the Solo® vibrating mesh nebulizer and the Wright® jet nebulizer

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster Cardio-Respiratory Research Lab, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No